CLINICAL TRIAL: NCT05953688
Title: A Proof-of-Concept, Randomized, Double-Masked Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Active Noninfectious Intermediate, Posterior, or Panuveitis (OPTYK-1)
Brief Title: POC Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Active Intermediate, Posterior, or Pan NIU
Acronym: OPTYK-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated based on interim efficacy data that did not meet the Sponsor's criteria.
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESK-001-014
Record Dates: First submitted 2023-06-29; First posted 2023-07-20 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Uveitis Posterior Non-Infectious; Uveitis, Intermediate; Noninfectious Panuveitis
MeSH Terms: conditions — Uveitis, Intermediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESK-001 Dose Level 1 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 2 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001

INTERVENTIONS:
Drug: ESK-001 — Oral tablet

SUMMARY:
This is a multi-center, randomized, double-masked, proof-of-concept study in patients with Active Noninfectious Intermediate, Posterior, or Panuveitis.

DETAILED DESCRIPTION:
This study will consist of a 2-week screening period (+7 days), 24-week treatment period, followed by a 24-week extension period, and a 4-week follow up period for a total of up to 55 weeks. Each participant will be randomized to receive one of two doses of ESK-001 daily for 24 weeks. Participants that do not meet the treatment failure criteria at Week 24 will continue into the extension period.

ELIGIBILITY:
Key Inclusion Criteria:

* Able and willing to provide consent
* Male and females, age 18 to 70 years
* Diagnosis of active noninfectious intermediate, posterior or panuveitis
* Must have active uveitis at Screening in at least one eye as defined by:

  1. Active inflammatory chorioretinal and/or inflammatory retinal vascular lesion or lesions, or
  2. ≥ 2+ VH in accordance with the NEI/SUN criteria
* Males and females must use highly effective methods of contraception for the entirety of the study

Key Exclusion Criteria:

* Diagnosis of infectious uveitis
* Has elevated intraocular pressures or severe glaucoma
* Positive for HIV, Hepatitis B or C or active or inadequately latent tuberculosis at screening
* Positive for syphilis at screening
* Patients with QTcF >450 msec (both males and females) at screening
* Known active malignancy or history of malignancy within the past 5 years
* History of chronic drug or alcohol abuse
* Live vaccines
* No planned ocular or any other surgery during the course of the study

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy between 2 ESK-001 treatment groups for the treatment of active NIU as measured by the proportion of patients failing treatment by Week 24 | 24 Weeks
  The proportion of patients failing treatment for active NIU by Week 24 between 2 ESK-001 treatment groups. Treatment failure is defined as a patient meeting at least 1 of the treatment failure criteria in at least 1 eye at Week 24.

SECONDARY OUTCOMES:
To compare the efficacy between 2 ESK-001 treatment groups for the treatment of active NIU as measured by the time to treatment failure on or after Week 24 | 24 Weeks
  Time to treatment failure on or after Week 24 between 2 ESK-001 treatment groups. Time to treatment failure is defined as time to the visit of the first treatment failure as defined per protocol. Median time to treatment failure in each treatment group will be reported and compared.
To assess the safety and tolerability of ESK-001 in patients with active NIU by comparing the incidence and proportion of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | Through study completion, up to 52 weeks
  Clinical and laboratory assessments including blood tests, ECGs, hematological measures and physical examinations throughout the study. The number and proportion of TEAEs, SAEs, AEs leading to study discontinuation, and AEs of greater than grade 3 severity will recorded per treatment group and across all groups.
To characterize the pharmacokinetics (PK) of ESK-001 (Cmax) | Through study completion, up to 48 weeks
  Plasma concentrations and PK parameters including steady-state maximum observed concentration (Cmax) for ESK-001 at Day 1, Week 24, and Week 48.
To characterize the pharmacokinetics (PK) of ESK-001 (Ctrough) | Through study completion, up to 48 weeks
  Plasma concentrations and PK parameters including steady-state trough observed plasma concentration (Ctrough) for ESK-001 at Week 24, and Week 48.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Investigator Site#1065, Beverly Hills, California
  - Investigator Site #1073, Los Angeles, California
  - Investigator Site #1072, Los Angeles, California
  - Investigator Site #1080, Palo Alto, California
  - Investigator Site #1079, Sacramento, California
  - Investigator Site#1068, Lakewood, Colorado
  - Investigator Site #1086, Oak Park, Illinois
  - Investigator Site #1085, Hagerstown, Maryland
  - Investigator Site #1069, Waltham, Massachusetts
  - Investigator Site #1076, Palisades Park, New Jersey
  - Investigator Site #1083, Durham, North Carolina
  - Investigator Site #1064, Erie, Pennsylvania
  - Investigator Site#1066, Nashville, Tennessee
  - Investigator Site #1084, Nashville, Tennessee
  - Investigator Site#1075, Bellaire, Texas
  - Investigator Site #1074, Katy, Texas
  - Investigator Site #1078, Plano, Texas

IPD SHARING:
Plan to Share IPD: No